CLINICAL TRIAL: NCT06527781
Title: A Phase 1a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of PD5K3 in Healthy Adult Volunteers
Brief Title: A Study of PD5K3 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-PK-PD5K3-14
Record Dates: First submitted 2024-07-19; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Lymphoblastic Leukemia, Acute; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: PD5K3 group and placebo control group are double-blinded, while the active comparator group is open-labeled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD5K3 group (Experimental): Eight subjects will be randomized to receive a single dose of PD5K3 in a double-blind fashion at each dose level.
  Interventions: Drug: PD5K3
- PD5K3 Placebo group (Placebo Comparator): Two subjects will be randomized to receive placebo in a double-blind fashion at each dose level.
  Interventions: Drug: Placebo
- Pegaspargase group (Active Comparator): Four subjects will receive a single dose of pegaspargase at the each dose level, and the dose of pegaspargase is the same with PD5K3. This group is open-labelled.
  Interventions: Drug: Pegaspargase

INTERVENTIONS:
Drug: PD5K3 — Six dose levels will be evaluated. intravenous injection
  Arms: PD5K3 group
Drug: Placebo — intravenous injection
  Arms: PD5K3 Placebo group
Drug: Pegaspargase — Six dose levels will be evaluated. intramuscular injection
  Other Names: Aiyang®
  Arms: Pegaspargase group

SUMMARY:
The main aim of this clinical trial is to assess the safety of PD5K3 in patients aged 18 to 65 years. The main questions it aims to answer are:

* Is PD5K3 safe in adult? Researchers will compare PD5K3 to an active comparator pegaspargase to see if PD5K3 is safe and active in human.

Participants will

* Receive a single dose injection of PD5K3, pegaspargase or placebo according to weight,
* Visit the clinic for assessment.

DETAILED DESCRIPTION:
This study is a first-in-human study, which is a single-center, randomized, placebo-controlled, double-blind, dose escalation, clinical study, aiming to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of PD5K3 in healthy adult volunteers, compared with pegaspargase at the same dose.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy male or female subjects;
2. Aged 18 to 65 years (inclusive);
3. The body mass index (BMI) in the range 18.0~28.0 kg/m^2 (inclusive);
4. Voluntarily participate and sign the informed consent form;
5. Be able to complete the trial in accordance with the protocol.

Exclusion Criteria:

1. Suffering from any diseases of the circulatory system, digestive system, urinary system, respiratory system, nervous system, endocrine system, reproductive system, etc. or any other diseases that can interfere with the test results;
2. Abnormal results with clinically significance of comprehensive physical examination, vital signs, laboratory tests (blood routine, blood biochemistry, seven coagulation items, urine routine, myocardial enzymes), 12-lead electrocardiogram, chest X-ray (anteroposterior), abdominal B-ultrasound (liver, gallbladder, pancreas, spleen and kidney);
3. Allergic constitution, including allergic to asparaginase;
4. Used PEGylated drugs in the past;
5. Fasting blood glucose ≥ 6.1mmol/L;
6. Have difficulty in venous blood collection, have a history of needle phobia or blood phobia, or have a known severe bleeding tendency;
7. Positive urine test for drug abuse;
8. Positive breath test for alcohol;
9. Smoke excessively (average > 5 cigarettes/day) within 3 months before screening or cannot stop using any tobacco products during the trial;
10. Drink excessively every day within 3 months before screening (male daily alcohol consumption exceeds 25g, such as 750 mL of beer, 250 mL of wine, or 75 mL of 38° liquor; female daily alcohol consumption exceeds 15g, such as 450 mL of beer, 150 mL of wine, or 50 mL of 38° liquor), or cannot abstain from alcohol during the trial;
11. Drink excessive amounts of tea, coffee or caffeinated beverages every day within 3 months before screening (more than 8 cups per day, 1 cup = 250 mL);
12. One or more positive tests for hepatitis B virus surface antigen, hepatitis C virus antibody, syphilis specific antibody, and human immunodeficiency virus antibody;
13. Female subjects are in lactation or have positive blood pregnancy test during the screening period or trial;
14. Undergone surgery within 3 months before screening or plan to undergo surgery during the trial;
15. Donated blood or lost more than 400 mL of blood within 3 months before screening (excluding menstrual bleeding);
16. Participated in any clinical trial as a subject within 3 months before screening;
17. Took any prescription drugs, over-the-counter drugs, health products, and any functional vitamins or Chinese herbal products within 28 days before administration;
18. The subject or his/her partner is unwilling to use one or more non-drug contraceptive measures (such as complete abstinence, condoms, contraceptive rings, ligation, etc.) for contraception during this trail or have a fertility plan within 6 months after the end of the study;
19. The investigator believes the subject would be unsuitable for participation in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse Events | up to 49 days
  To evaluate the adverse events as characterized by type, frequency, severity as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, timing, seriousness, and relationship to study therapy after administration.

SECONDARY OUTCOMES:
The Area Under the Curve from dosing to the time of the last measured concentration (AUC0-t) | up to 49 days
  Pharmacokinetic parameter
Maximum plasma concentration (Cmax) | up to 49 days
  Pharmacokinetic parameter
The half-life (t1/2) | up to 49 days
  Pharmacokinetic parameter
Compare the plasma asparaginase activity between the PD5K3 and pegaspargase groups | up to 49 days
  Plasma asparaginase activities are determined by a validated enzymatic spectrophotometric assay, and the results are reported in IU/mL. In the assay, asparaginase hydrolyzes asparagine to generate aspartic acid, which can be detected colorimetrically using a coupled enzymatic reaction.
Compare the plasma asparagine concentration between the PD5K3 and pegaspargase groups | up to 49 days
  Plasma asparagine concentration as a pharmacodynamic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangshu, China